CLINICAL TRIAL: NCT06819670
Title: A Multicenter Pilot Clinical Trial to Prevent Infantile Spasms Relapse
Brief Title: A Study to Prevent Infantile Spasms Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Pediatric Epilepsy Research Foundation (Unknown)
Responsible Party: Principal Investigator, Shaun Hussain, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-001710; 20224426 (Other Grant/Funding Number: Pediatric Epilepsy Research Foundation)
Record Dates: First submitted 2025-01-29; First posted 2025-02-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Infantile Spasms; Infantile Epileptic Spasms Syndrome; West Syndrome
Keywords: Relapse; Infantile Spasms; Prednisolone
MeSH Terms: conditions — Spasms, Infantile; Recurrence | interventions — Prednisolone; Famotidine

STUDY DESIGN:
Intervention Model Description: Prednisolone (1 mg/kg/day) or placebo AND famotidine (1 mg/kg/day) or placebo. Both medications will be administered daily for 4 months, followed by a 1-month taper
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose prednisolone (Active Comparator): Prednisolone and famotidine.
  Interventions: Drug: Prednisolone; Drug: Famotidine
- Placebo (Placebo Comparator): Placebo (prednisolone) and placebo (famotidine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — active drug
  Arms: Low-dose prednisolone
Drug: Famotidine — active drug
  Arms: Low-dose prednisolone
Drug: Placebo — non-active drug
  Arms: Placebo

SUMMARY:
After initially successful treatment, many children with infantile spasms unfortunately have a relapse, and relapse is linked to poor long-term outcomes such as autism and other forms of epilepsy. The aim of this study is to determine if treatment with low-dose prednisolone is safe, well tolerated, and effective in reducing the risk of relapse.

DETAILED DESCRIPTION:
In this study, the investigators will enroll infants who have responded to standard therapy for treatment of Infantile Epileptic Spasms Syndrome (IESS). Patients will be randomized to receive either low-dose prednsiolone or placebo for 4 months. During the first 7 months, patients will be evaluated monthly, with clinic visits and electroencephalography (EEG). Patients will then return for a final visit at age 2 years. Key outcomes will be determination of IESS relapse, emergence of other types of seizures/epilepsy, and evaluation of developmental/behavioral status at age 2 years. We will attempt to determine whether or not the prednisolone intervention reduces the risk of any adverse outcome, but this may not be possible given the study design. We will also evaluate the feasibility of the intervention, study procedures, and recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 to 18 months, inclusive
2. Clinical diagnosis of infantile spasms syndrome, with EEG-confirmed complete response to standard treatment (prednisolone, ACTH, and/or vigabatrin)

Exclusion Criteria:

1. Presence of clinically significant hypertension, infection, or any other diagnosis which poses unreasonable risk in the setting of extended corticosteroid therapy, in the view of the study physician
2. Exposure to any artisanal cannabinoid product within 14 days of screening
3. Ongoing therapy with the ketogenic diet
4. Implantation of a vagal nerve stimulator within 3 months of screening, or any change in stimulation parameters within 1 month of screening
5. Treatment of IESS via epilepsy surgery

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From enrollment to 5-month visit.
  The investigators will tabulate of adverse events and determine whether any adverse event is associated with prednisolone treatment during the first 5 months of the study.
Incidence of epileptic spasms relapse | From enrollment to last evaluation at age 2 years
  The investigators will record whether or not study participant experience a relapse of epileptic spasms during the study. Relapse is classified as present or absent and based on interpretation of EEG.

SECONDARY OUTCOMES:
Incidence of autism spectrum disorder | From enrollment to last evaluation at age 2 years
  At the final study visit, the investigators will use DSM-V criteria to determine if study participants fulfill diagnostic criteria for autism spectrum disorder.
Developmental/Behavioral Level | From enrollment to last evaluation at age 2 years
  At the final study visit at age 2 years, the investigators will measure adaptive behavior using the Vineland-3 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun A. Hussain, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be shared with other researchers upon reasonable request, after publication of results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be shared upon reasonable request after publication of study results.
Access Criteria: Deidentified patient data, study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code.

REFERENCES:
- [Background] Hussain SA. Treatment of infantile spasms. Epilepsia Open. 2018 Oct 23;3(Suppl Suppl 2):143-154. doi: 10.1002/epi4.12264. eCollection 2018 Dec. PMID 30564773
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30564773/